CLINICAL TRIAL: NCT00000972
Title: A Phase I Clinical Trial to Evaluate: Part A. The Safety of MTP-PE/MF59 Adjuvant Emulsion. Part B. The Safety and Immunogenicity of Env 2-3, a Yeast Derived Recombinant Envelope Protein of Human Immunodeficiency Virus-1, in Combination With MTP-PE/MF59
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Biocine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Prevention
Other Study IDs: AVEG 005A/B; 10546 (Registry Identifier: DAIDS ES Registry Number); 10547 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Vaccines, Synthetic; Drug Evaluation; Adjuvants, Immunologic; AIDS Vaccines; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: MTP-PE/MF59
Biological: Env 2-3

SUMMARY:
To evaluate the safety of a fixed antigen dose with an increasing dose of adjuvant (MTP-PE/MF59, a substance to enhance the immune response to vaccine) in volunteers. To evaluate local and systemic reactions (Part A). To determine the safety and immunogenicity of Env 2-3 in combination with MTP-PE/MF59 in volunteers (Part B). The vaccine Env 2-3 is created from one of the viral proteins that make up HIV called envelope glycoprotein gp120. A problem with many immunogens, including candidate HIV vaccines, is that they may evoke relatively weak immune responses, particularly in humans and in nonhuman primates. Thus, there is considerable interest in the development of "adjuvants" (substances that augment immune responses to vaccines). MTP-PE/MF59 is an adjuvant that appears to be particularly promising, and is selected for the studies with this HIV vaccine candidate.

DETAILED DESCRIPTION:
The vaccine Env 2-3 is created from one of the viral proteins that make up HIV called envelope glycoprotein gp120. A problem with many immunogens, including candidate HIV vaccines, is that they may evoke relatively weak immune responses, particularly in humans and in nonhuman primates. Thus, there is considerable interest in the development of "adjuvants" (substances that augment immune responses to vaccines). MTP-PE/MF59 is an adjuvant that appears to be particularly promising, and is selected for the studies with this HIV vaccine candidate.

This study is being conducted in two parts: Part A examines the safety of the adjuvant MTP-PE/MF59 alone; Part B examines the safety and immunogenicity of Env 2-3 in combination with MTP-PE/MF59. In Part A, three volunteers receive MTP-PE/MF59, and one volunteer receives emulsion alone at each dose level. Initiation of each dose level is separated by at least 72 hours. Doses of adjuvant emulsion are administered at day 0 and day 30 for the highest tolerated dose. If significant reactions are encountered, additional subjects may be studied at lower doses. In Part B, six doses of MTP-PE adjuvant (0, 5, 10, 25, 50, or 100 mcg) in the MF59 emulsion are studied. Six volunteers receive Env 2-3/MTP-PE/MF59 and two receive MTP-PE/MF59 alone at each dose level. There is a minimum 1-week interval between dose escalations. Per amendment, volunteers may receive an additional dose of Env 2-3 or placebo in MF59 emulsion only, administered 12-18 months post initial inoculation.

ELIGIBILITY:
Inclusion Criteria

Volunteers are:

* Normal, healthy adults (by history and physical examination) who fully comprehend the purpose and details of the study.

Part A:

* Available for 60 days.

Part B:

* Available for 1 year of follow-up.

Exclusion Criteria

Co-existing Condition:

Volunteers with the following conditions or symptoms are excluded: Part B:

* Positive syphilis serology (such as VDRL) unless positive test is due to a documented clinical event that occurred and was treated 5 or more years prior to enrollment.

Circulating hepatitis B antigenemia.

-

Volunteers with the following are excluded:

* History of immunodeficiency, chronic illness, autoimmune disease.
* Evidence of depression or under treatment for psychiatric problems during the past year.

Prior Medication:

Excluded:

* Immunosuppressive medications.

Prior Treatment:

Excluded: Part B:

* Blood transfusion or cryoprecipitates within the past 6 months.

Risk Behavior: Excluded: Part B: Identifiable high-risk behavior for HIV infection, including:

* history of intravenous drug use; syphilis, gonorrhea, or any other sexually transmitted diseases (including chlamydia or pelvic inflammatory disease) in the last 6 months; more than two sexual partners, or sexual contact with a high-risk partner, in the preceding 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Study Completion 1992-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolin R, Study Chair
Locations (3):
- United States (3):
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Evans TG, Fitzgerald T, Gibbons DC, Keefer MC, Soucier H. Th1/Th2 cytokine responses following HIV-1 immunization in seronegative volunteers. The AIDS Vaccine Evaluation Group. Clin Exp Immunol. 1998 Feb;111(2):243-50. doi: 10.1046/j.1365-2249.1998.00486.x. PMID 9486388
- [Background] Keefer MC, Graham BS, McElrath MJ, Matthews TJ, Stablein DM, Corey L, Wright PF, Lawrence D, Fast PE, Weinhold K, Hsieh RH, Chernoff D, Dekker C, Dolin R. Safety and immunogenicity of Env 2-3, a human immunodeficiency virus type 1 candidate vaccine, in combination with a novel adjuvant, MTP-PE/MF59. NIAID AIDS Vaccine Evaluation Group. AIDS Res Hum Retroviruses. 1996 May 20;12(8):683-93. doi: 10.1089/aid.1996.12.683. PMID 8744579